

# FMHS RESEARCH ETHICS COMMITTEE (REC) Ethics Application Form

# ONLY FULLY SIGNED (electronic) TYPE-WRITTEN APPLICATIONS WILL BE ACCEPTED, BY EMAIL or SHARED via OneDrive

Please complete this combined Form/Protocol template if your research study is **using qualitative**, **quantitative** or mixed or other methodology involving people and their data.

| STUDY DETAILS | | | |
|---|---|---|---|
| Full study title | Understanding the impacts and experiences of children of | urrently ex | periencing |
| | parental imprisonment | | |
| Short title/Acronym | IECPI | | |
| FMHS REC reference | | | |
| Date and version number | Version 1.0: 16.04.2025 | | |
| Principal Investigator | Dr Elizabeth Paddock, Assistant Professor in Forensic Psy<br>Medicine & Health Sciences | chology, Fa | culty of |
| University email contact | elizabeth.paddock@nottingham.ac.uk | | |
| Student (if applicable) | Miss Kyra Wardle, DForenPsy, Faculty of Medicine & Hea | ılth Science | S |
| University email contact | kyra.wardle@nottingham.ac.uk | | |
| University telephone contact | | | |
| Medically qualified/Healthcare professional collaborator (licensed doctor/registered nurse/Psychologist) | N/A | | |
| Sponsor | The University of Nottingham | | |
| Funder | None | | |
| Is this project a Collaboration Is there an agreement in pla | | ☐ Yes<br>☐ Yes | ⊠ No<br>⊠ No |
| If yes to either of above pleas | se give more details here | | |
| Will you submit or have you | u submitted this study to another ethics committee? | ☐ Yes | ⊠ No |
| | r this research are required (e.g. from other universities' eth<br>tutional Review Boards) please include with the application | | |

| Declaration of any | None |
|---|---|
| conflicts of interest | |
| DBS Check | Enhanced DBS completed as part of full-time role. Information available upon |
| | request. |
| Do you have a Data | The University expects a data management plan to be in place before a |
| Management Plan? | research project commences. Please see appendices. |
| | For further details see: <u>Digital Research</u> : |
| Confidentiality statement | This document contains confidential information that must not be disclosed to |
| | anyone other than the authorised individuals from the University of |
| | Nottingham, the Investigator Team and members of the Research Ethics |
| | Committee unless authorised to do so. |

| RESEARCH TEAM | |
|---|---|
| Principal investigator (PI)/Researcher title, | Kyra Wardle |
| name, Job title | DForenPsy Student |
| | Trainee Forensic Psychologist |
| | Lead Researcher |
| Research Group | School of Medicine |
| Department/institute/School | Centre for Forensic and Family Psychology |
| Role in study | Lead Researcher |
| Training/qualification in Research Integrity | BSc Psychology Degree 2020 (2:1). Dissertation published. |
| and research ethics and experience relevant | MSc Forensic Psychology and Mental Health 2022 |
| to the Proposed Research Activities | (Distinction). Dissertation currently editing for publication. |
| | DForenPsy Forensic Psychology (current) |
| Principal investigator (PI)/Researcher title, | Dr Elizabeth Paddock |
| name, Job title | HCPC Registered Practitioner Psychologist |
| Doctorate in Forensic Psychology Course Director | |
| Research Group | School of Medicine |
| Department/institute/School | Centre for Forensic and Family Psychology |
| Role in study | Research Supervisor |
| Training/qualification in Research Integrity | |
| and research ethics and experience relevant | |
| to the Proposed Research Activities | |

# **TABLE OF CONTENTS**

# Contents

| 1. TABLE OF CONTENTS | 3 |
|---|---|
| 2. LAY SUMMARY | 4 |
| 3. SYNOPSIS | 5 |
| 4. ABBREVIATIONS | 11 |
| 5. BACKGROUND AND RATIONALE | 12 |
| 6. AIM / RESEARCH QUESTIONS / OBJECTIVES | 12 |
| 7. STUDY DESIGN | 12 |
| 8. PARTICIPANTS | 18 |
| 9. ETHICAL CONSIDERATIONS AND PARTICIPANT AND RESEARCH | IER SAFETY24 |
| 10. DATA MANAGEMENT SUMMARY | 27 |
| 11. STUDY MONITORING AND OVERSIGHT | 29 |
| 12. ETHICAL AND REGULATORY CONSIDERATIONS | 29 |
| 13. INSURANCE AND INDEMNITY | 29 |
| 14. DISSEMINATION AND FEEDBACK OF STUDY OUTCOMES | 30 |
| 15. REFERENCES | 30 |
| 16. DECLARATIONS AND SIGNATURES | 32 |
| 17. AMENDMENT HISTORYE | rror! Bookmark not defined |
| 18. Useful links: | 33 |
| 19. Check List | 34 |

#### LAY SUMMARY

It is estimated that over 100,000 children in England and Wales are separated from their parents due to parental imprisonment (Aebi et al., 2023), now recognised as an adverse childhood experience that can have multifaceted challenges for the families and children associated (ACEs; Felitti et al., 1998).

Separation from a parent under any circumstance can be experienced by a child as distressing and traumatic, however, researchers have likened the experience and impacts of parental imprisonment to losing a parent to death or divorce (Lowenstein, 1986). Parental imprisonment is an ambiguous loss for a child, and is often characterised by the sudden loss of an attachment figure, however, this is coupled with stigmatisation and discrimination associated with offending. A considerable research base focusing on the non-offending partners has highlighted that the imprisonment of a loved one can result in experiences of disenfranchised grief, stigmatisation, and symptoms of trauma (Duncan et al., 2022). It is possible that children may internalise the stigma attached to having a parent in prison, or the offence committed, which can result in low self-esteem, self-worth, and increased isolation (McGinley et al., 2018), however, there remains scarce research focusing on children's experiences of parental separation by imprisonment, and how they make sense of this.

Utilising quantitative methods, research has found that parental imprisonment is associated with increased rates of mental health problems, major depression and attention disorders in comparison to the general population (Murray & Farrington, 2007). Similarly, research has found that following parental imprisonment, children experienced depression, difficulties attending and concentration in school, chronic sleeplessness, loneliness, increased substance misuse, and financial challenges (Arditti, 2016; Murray et al., 2012; Sack et al. 1987 as cited in Parke and Clarke-Stewart 2001). In comparison to the general population, prisoners are also more likely to have experienced socioeconomic disadvantages, mental health problems, and marital difficulties, which are all found to be risk factors for mental health problems in children. Bulow (2014) supported this, suggesting that parental imprisonment has a disproportionate impact on children associated as a result of imprisonment magnifying existing social and economic disadvantages. It is therefore possible that pre-existing factors to parental imprisonment impact on child outcomes, and that parental imprisonment acts as a catalyst (Dobbie et al., 2019).

Despite a body of quantitative research attempting to understand the impacts of parental imprisonment on child outcomes (Murray, 2005), much is still unknown of a child's own experiences of parental imprisonment. An emerging evidence base has utilised qualitative methods with children, finding contrasting results. In Noel and Hoeben's (2022) research, children reported that parental imprisonment was a negative experience resulting in financial challenges, lack of support, and reduced academic opportunities, whilst others shared that parental imprisonment was a positive experience. Similarly, Muhammed (2011) in their study of interviews with children between 7 and 18 years with a parent in prison, found that the impacts described by children were different to how these were described by other's surrounding the child.

It is clear from the evidence base that children impacted by parental imprisonment are not a homogenous group, and research is required to understand the experiences of parental imprisonment on a child, within the context of individual risk and protective factors.

This research aims to understand the impacts, experiences, and support needs of children who are aged 16 years and above, currently experiencing parental imprisonment from their own perspective, and from the perspective of their non-offending parent/caregiver/guardian and a professional. This research will adopt a case study design. Semi-structured interviews will be conducted with the child experiencing parental imprisonment, and the non-offending parent or caregiver. This research will also aim to recruit a professional working with the young person or family during parental imprisonment. This will be analysed interpretative phenomenological analysis.

#### **SYNOPSIS**

| | DForenPsy Student project |
|---|---|
| Type of Project | Qualitative methodology |
| | Study involving children (above 16 years old). |
| List all sites where | |
| this study will be | Online semi-structured interviews conducted via Microsoft Teams |
| conducted | |
| Age range of study participants | 16 years and above. |
| | This research aims to utilise a case study format. This research will aim to recruit a |
| | minimum of one case study, inclusive of a child (referring to an individual above 16 |
| | years old, whose parent has been imprisoned) currently experiencing parental |
| Sample size and | imprisonment, and their non-offending parent/caregiver or guardian. It is also hoped |
| groups | that this research will recruit one professional working with the child or family member. |
| | This research will therefore recruit a minimum of one case study (minimum of two |
| | participants per case study), and a maximum of five case studies. |
| | Participants will be recruited through voluntary purposive sampling. The research will |
| Study Participants, | be advertised on several social media platforms (including LinkedIn, Twitter, and |
| including sampling | Reddit), and organisational and charitable websites that work with families of those |
| strategy | convicted of offences (including Children Heard and Seen, Safer Lives, Prison Advice |
| | Care Trust; PACT). |
| Planned study | |
| duration | 6 months |
| Anticipated start date | Projected start date for study: following Ethics approval. |

| | Projected start date for recruitment and o | data collection: following Ethics approval. |
|---|---|---|
| Anticipated end date | Projected end date: 01/01/2026 | |
| | Aim/Research Question | Objectives |
| Aim/Research Questions/Objectives | What are the impacts and experiences of children currently experiencing parental imprisonment? | To understand the impacts and experiences of children currently experiencing parental |
| | imprisonment? 2. What are the protective factors to parental imprisonment described by children currently experiencing this? | <ul> <li>imprisonment.</li> <li>2. To understand the support needs of children experiencing parental imprisonment.</li> <li>3. To know if the impacts,</li> </ul> |
| | <ul> <li>3. How do the non-offending parents/carers/guardians understand the impact and experiences to children of having a parent in prison?</li> <li>4. What are the support needs of children experiencing parental imprisonment?</li> </ul> | experiences and support needs of children experiencing parental imprisonment are understood by caring figures. |
| Study Design, including methodology | parental imprisonment, and their non-orecruited. This research will also aim to refamily during parental imprisonment. Adult participants Adult participants refer to the non-offeryears old. The research will consist of one and the lead researcher. Participant computer/laptop or phone to attend the date and time of the interview will be schedard participant. The participants will be as feel is safe and confidential. The interview | n, whereby one child currently experiencing offending parent/caregiver/guardian will be ecruit a professional working with the child or ending parent/caregiver/guardian above 18 e-to-one interviews between the participants interview via Microsoft Teams or Zoom. The eduled at conveniency for both the researcher sked to complete the interview in a place they ew will be semi-structured which will consist to take approximately 1 hour. The interview |

# Child participants

The research will consist of one-to-one interviews between the participants and the lead researcher. The research refers to children participants as individuals who are above 16 years old, and have a parent currently in prison. The children participants will be interviewed one-to-one. Participants will be asked to use their personal computer/laptop or phone to attend the interview via Microsoft Teams or Zoom. The date and time of the interview will be scheduled at conveniency for both the researcher and participant. The interview will be semi-structured which will consist open questions and this is anticipated to take approximately 1 hour. The interview schedule is attached. The interview will also utilise a timeline activity to promote engagement and discussion.

# **Professional participants**

This refers to professionals working with the young person or family during parental imprisonment. The research will consist of one-to-one interviews between the participants and the lead researcher. Participants will be asked to use their personal computer/laptop or phone to attend the interview via Microsoft Teams or Zoom. The date and time of the interview will be scheduled at conveniency for both the researcher and participant. The participants will be asked to complete the interview in a place they feel is safe and confidential. The interview will be semi-structured which will consist open questions and this is anticipated to take approximately 1 hour. The interview schedule is attached.

# **Analysis**

This research will be analysed using interpretative phenomenological analysis (IPA; Smith et al., 2022). IPA is concerned with phenomenology, the study of subjective experience which aims to understand how people make sense of major life events. The current research will adopt an idiographic stance, that is interested in an individual's experience and how they make sense of it. This research will also adopt a contextualist stance, which understands that stories can access' participants perceptions and understanding of personal experiences, but that these are shaped by and embedded in the participants social context (Moller et al., 2021).

This research focuses on the children's experiences and impacts of parental imprisonment. Whilst IPA studies traditionally collect data from a sample with a shared experience, this research will also recruit the non-offending parents and professionals to provide their perspective of the child's experiences and impacts. In the current

study, the child's voices will be prioritised and analysed first and separate to that of adult and professional data.

The analysis will adhere to the principles of interpretative phenomenological analysis as outlined by Smith et al., (2022). Careful consideration will be given to the order in which data is analysed. As this research focuses on the children's voices and experiences, interviews completed with children will be analysed first to ensure that analysis of adult and professional data does not influence the interpretation.

# Purpose of tool to be used in this study

The semi-structured interviews will be conducted using Microsoft Teams, which has been identified as the most appropriate online platform for participation.

Additionally, child interviews will be supported using a timeline activity. Timelines have been used in previous qualitative research with children, and has been cited to be a useful resource in facilitating conversation, focusing a participant's attention and recollection of events (King et al., 2019; Smith & Paddock, 2024). Furthermore, the use of timeline activities have been suggested to be helpful in building rapport with participants, mediating power imbalance, anticipated when working with children, and minimising distress that may be experienced by the participant when talking about difficult and distressing topics due to the refocus of their attention (Kolar et al., 2015).

# Potential problems posing a particular risk to participant and researcher.

This research focuses upon personal experiences of children, and the non-offending parent/caregiver/guardian currently experiencing parental imprisonment. There is potential for this to cause for psychological distress given that this research focuses upon their own personal experiences.

The research will take several precautions to minimise these risks:

# **Participant Recruitment:**

- Participants will be provided with a full and comprehensive outline of the proposed study and what the questions might elicit. Please see appendices.
- The current research will be advertised on online platforms, local services, and by non-governmental organisations. Participants will be provided with services whom they can contact for support.

# Preliminary discussion with researcher:

 Prior to partaking in this research, it will be requested that the participants attend a preliminary discussion with the researcher (preferably via call on Microsoft Teams, but also via email exchange). During this, the participant will be encouraged to ask any questions they have about their involvement in this research. It will also seek to understand:

- o Participants' current wellbeing and mental health.
- The child participants' understanding of their parent's imprisonment and offence.
- Ascertain if there is a professional that knows and works closely with the family/ child participant that can participate in the research (if there are, they will also be offered the same preliminary discussion as the adult participant).
- During the preliminary discussion with the child participant, they will be
  offered an opportunity to request the non-offending parent to be present
  during the interview.

In the preliminary discussions with the adult, child, and professional participants, the researcher will explain the current project:

- The researcher will outline and explain the ability to withdraw from the study at any time without reason up until two weeks after the interview date.
- The researcher will explain the themes and types of questions which will be asked within the interview.
- The researcher will provide a warning to the participant that this research topic
  and area is sensitive and that if participants feel they are in a vulnerable place
  in their life, not doing too well and have any doubt that they would feel unable
  to cope, it will be advised that they do not participate in this research.
- If participants who initially wanted to participate in this research, and after the
  preliminary discussion do not want to participate, the debrief form will still be
  provided.

# **Participant Interview**

- At the time of the interview, the researcher will once again explain and outline the study and sensitive nature of such.
- It will be reiterated that if they feel they are in a vulnerable place in their life, not doing too well or feel unable to cope, they will be advised to not partake in the study.
- Participants will be reminded that throughout the interview they can break at any time and also withdraw, without the need for a reason.

- If participants would like to withdraw during the interview, the debrief form will still be provided.
- Once the interview begins, the first couple of questions will be asked and the
  researcher will check in with the participant regarding how they are feeling and
  if they would like to continue.
- A mandatory break will be provided halfway through the interview schedule.
- The adult interview will be conducted prior to the child interview in order for the lead researcher to understand context.
- Child interviews will be supported using a timeline activity. Timelines have been used in previous qualitative research with children, and has been cited to be a useful resource in facilitating conversation, focusing a participant's attention and recollection of events (King et al., 2019; Smith & Paddock, 2024). Furthermore, the use of timeline activities have been suggested to be helpful in building rapport with participants, mediating power imbalance, anticipated when working with children, and minimising distress that may be experienced by the participant when talking about difficult and distressing topics due to the refocus of their attention (Kolar et al., 2015).

# After interviews

 After each interview, or at any point of withdrawal, participants will be provided with information for access to support services, both specific and general and will be encouraged to access these.

# **ABBREVIATIONS**

| DMP | Data Management Plan |
|---------|-----------------------------------------------------------|
| FMHS | Faculty of Medicine & Health Sciences |
| GCP | Good Clinical Practice |
| GP | General Practitioner |
| ICF | Informed Consent Form |
| PI | Principal Investigator |
| PIS | Participant Information Sheet |
| SOP | Standard Operating Procedure |
| UoN | University of Nottingham |
| REC | Research Ethics Committee |
| PI | Parental Imprisonment |
| ACES-IQ | Adverse Childhood Experiences International Questionnaire |
| SC | Story Completion |

#### **BACKGROUND AND RATIONALE**

#### AIM / RESEARCH QUESTIONS / OBJECTIVES

# Aim/Research questions

- What are the impacts and experiences of children currently experiencing parental imprisonment?
- 2. What are the protective factors to parental imprisonment described by children currently experiencing this?
- 3. How do the non-offending parents/carers/guardians understand the impact and experiences to children of having a parent in prison?
- 4. What are the support needs of children experiencing parental imprisonment?

# **Objectives**

- 1. To understand the impacts and experiences of children currently experiencing parental imprisonment.
- 2. To understand the support needs of children experiencing parental imprisonment.
- 3. To know if the impacts, experiences and support needs of children experiencing parental imprisonment are understood by caring figures.

#### STUDY DESIGN

# Methodology

#### **Case Study Design**

# **Adult Interview**

The adult participant refers to the non-offending parent/ caregiver/ or guardian of the child participant. This research will consist of one-to-one semi-structured interviews between the adult participant and the lead researcher. Participants will be asked to use their personal computer/laptop or phone to attend the interview via Microsoft Teams or Zoom. The date and time of the interview will be scheduled at conveniency for both the



researcher and participant. The participants will be asked to complete the interview in a place they feel is safe and confidential. The interview will be semi-structured which will consist open questions and this is anticipated to take approximately 1 hour.

# Child Interview

This research will consist of semi-structured interviews between the child participant and the lead researcher.

Participants will be asked to use their personal computer/laptop or phone to attend the interview via Microsoft

Teams or Zoom. The date and time of the interview will be scheduled at conveniency for both the researcher and participant. The participants will be asked to complete the interview in a place they feel is safe and confidential. The interview will be semi-structured which will consist open questions and this is anticipated to take approximately 1 hour.

Additionally, the interview schedule will be supported using a timeline activity. Timelines have been used in previous qualitative research with children, and has been cited to be a useful resource in facilitating conversation, focusing a participant's attention and recollection of events (King et al., 2019; Smith & Paddock, 2024). Furthermore, the use of timeline activities have been suggested to be helpful in building rapport with participants, mediating power imbalance, anticipated when working with children, and minimising distress that may be experienced by the participant when talking about difficult and distressing topics due to the refocus of their attention (Kolar et al., 2015).

# **Professional Interview**

The professional interview will consist of one-to-one semi-structured interviews between the professional participant and the lead researcher. The professional interview will be selected by the non-offending parent/carer/guardian participant. The non-offending parent/carer/guardian participant or child participant will be asked to forward the research poster to the professional who will then have the opportunity to contact the research if they want to participate in the current research.

# **Analysis**

This research will be analysed using interpretative phenomenological analysis (IPA; Smith et al., 2022). IPA is concerned with phenomenology, the study of subjective experience which aims to understand how people make sense of major life events. The current research will adopt an idiographic stance, that is interested in an individual's experience and how they make sense of it. This research will also adopt a contextualist stance, which understands that stories can access' participants perceptions and understanding of personal experiences, but that these are shaped by and embedded in the participants social context (Moller et al., 2021). The child interviews will be analysed first and separate to that of the adult and professional interview data.

# **Sampling Strategy**

The non-offending parent/caregiver guardian and the child participant will be recruited through voluntary purposive sampling. The research will be advertised on several social media platforms (including LinkedIn, Twitter, and Reddit), and organisational and charitable websites that work with families of those convicted of offences (including but not limited to Children Heard and Seen, Safer Lives, and Prison Advice Care Trust).

The professional participant will be recruited via opportunity sampling. The non-offending parent/caregiver guardian participant will be encouraged to share the research poster with a professional that works with the family/young person who will then have the option to volunteer to partake in this research.

#### **Methods of Data Collection**

The research will be advertised on online platforms using a poster. This research will be advertised on online platforms such as LinkedIn and Mumsnet. It will also be advertised by non-governmental organisations that work with families of prisoners, or those involved with the Criminal Justice System (for example, Lucy Faithfull Foundation and Prison Advice Care Trust). At the point of the adult or child participant contacting the researcher to partake in this research, the participant will ask for this research to be shared with either the adult or child interview. It will be requested that both the adult and child participants partake in this research. The adult and child participant will be asked to volunteer for the research, and to provide consent.

The research will utilise a case study design which aims to recruit a child currently experiencing parental imprisonment, and their non-offending parent/guardian/caregiver. This will research will also aim to recruit a professional working with the child/family during parental imprisonment, though not essential. This research will utilise qualitative methods via semi-structured interviews.

The interviews will be conducted remotely via Microsoft Teams. The participants will be asked if they have access to these sites, a personal computer and are able to be in a private and quiet space during the interview. The researcher will also be in a quiet and private space. The interviews will be conducted via Teams and will be recorded using this function on Teams. The interviews will also be transcribed live using the online transcribing feature of Teams. This will be on a password protected laptop. The audio file will be password protected and saved as the participant number so that this is not identifiable. Demographics that are recorded will be stored separately, password protected and saved so that it is not identifiable. Once interviews are completed, the researcher will go through the recording and transcription to ensure that they are congruent. The transcription document will be password protected saved and stored securely on password protected device. During transcription, any identifiable information will be pseudonymised whereby they will be changed. Pseudonyms will be used in replacement of any identifiable information. This research will also utilise NVivo in the data analysis, a qualitative software which has been identified as adding validity to qualitative research (bringer et al., 2004). The data inputted into this software will be the pseudonymised formatted transcribed data.

This research cannot be completely anonymous as in the dissemination of findings, direct quotes may be taken from the pseudonymised interviews. However, any information included will not be identifiable to an individual (including their name, geographical place etc). Furthermore, any direct quotes used will focus on their experiences rather than the individual themselves, and this will be referred to using a generated pseudonymised name.

The adult, child, and professional interviews will be analysed using Interpretative Thematic Analysis separately to each other.

#### **Adult Interview**

Demographic information will be sought from non-offending parent/ guardian/ caregiver participants, including:

- 1. Age
- 2. Gender
- 3. Relationship to the child and individual in prison
- 4. Gender of parent imprisoned
- 5. Age their child experienced parental imprisonment
- 6. Offence type
- 7. Sentence Length
- 8. What area they currently reside in
- 9. What area the prison is based/distance between current residence and prison

The adult interview will be guided by a semi-structured interview schedule.

# **Child Interview**

Demographic information will be sought from the child participant, including:

- 10. Age
- 11. Gender
- 12. Age they experienced parental imprisonment
- 13. Relationship to the parent in prison
- 14. Age experienced parental imprisonment
- 15. Offence type
- 16. Sentence Length
- 17. What area they currently reside in
- 18. What area the prison is based/distance between current residence and prison

The child interview will be guided by a semi-structured interview schedule and utilise a timeline activity.

# **Professional Interview**

Demographic information will be sought from the child participant, including:

- 19. Age
- 20. Gender
- 21. Relationship to the child and individual in prison
- 22. Job and support they provide to the child/family

The professional interview will be guided by a semi-structured interview schedule.

# **Study Sequence and Duration**



#### **Data Collection:**

- 1. The research will be advertised on social media platforms and by charitable or non-governmental organisations.
- 2. Participants will be directed to contact the researcher to partake in this research.
- 3. Participants will be requested to complete a short demographic questionnaire, provided with an information sheet, and asked to share information about the research with the adult or child participant.
- 4. The participants will then be offered an opportunity to meet with the lead researcher for a preliminary discussion about this research, what to expect, and ask any further they question they have. This preliminary discussion can take place via Email, or over Microsoft Teams. Participants will be provided with a consent sheet.
- 5. Following the adult and child participant interview, participants will be invited to share the research poster with a professional that works with the child or family to partake in the current research who can volunteer to partake.
- 6. The professional participant will then be provided with information regarding the research and invited to a preliminary discussion. The professional participant will be invited for an interview with the researcher, following which they will be provided with information regarding support and debrief.

The research will be advertised until for approximately 6 months. The research aims to recruit a minimum of one case study. 'One case study' refers to at least one child participants and one non-offending parent/carer/guardian participant.

# **Data Analysis**

- 1. The interviews will be recorded on Microsoft Teams and transcription services used. The interviews will then be pseudonymised and any identifiable information will be destroyed.
- 2. The transcribed interviews will then be uploaded to NVivo for analysis and following all data collection.
- 3. This research will be analysed using interpretative phenomenological analysis (IPA; Smith et al., 2022). IPA is concerned with phenomenology, the study of subjective experience which aims to understand how people make sense of major life events.
- 4. The analysis will adhere to the principles of interpretative phenomenological analysis as outlined by Smith et al., (2022). Careful consideration will be given to the order in which data is analysed. As this research focuses on the children's voices and experiences, interviews completed with children will be analysed first to ensure that analysis of adult and professional data does not influence the interpretation.
- 5. The child interviews will be analysed first and separate to that of the adult and professional interview data.

# Number of participants & group allocations

This research utilises a case study design, that is inclusive of a child participant currently experiencing parental imprisonment and one adult participant whom is the non-offending parent/guardian/caregiver to the child. The research will also aim to recruit a professional working with the child or family impacted by parental imprisonment as part of the case study design, though not essential.

This research utilises IPA to understand an individual's major life event, and how they make sense of this. As such, IPA requires a small sample size. This research will recruit at least one case study, and a maximum of ten case studies.

# **Methods of Data Analysis**

# Quantitative

The quantitative data collected will primarily be collecting demographic data.

# Qualitative

Following qualitative data collection, the data will be pseudonymised and saved on a home-based password protected laptop. This research will be analysed using interpretative phenomenological analysis (IPA; Smith et al., 2022). IPA is concerned with phenomenology, the study of subjective experience which aims to understand how people make sense of major life events. The current research will adopt an idiographic stance, that is interested in an individual's experience and how they make sense of it. This research will also adopt a contextualist stance, which understands that stories can access' participants perceptions and understanding of personal experiences, but that these are shaped by and embedded in the participants social context (Moller et al., 2021).

The analysis will adhere to the principles of interpretative phenomenological analysis as outlined by Smith et al., (2022). Careful consideration will be given to the order in which data is analysed. As this research focuses on the children's voices and experiences, interviews completed with children will be analysed first to ensure that analysis of adult and professional data does not influence the interpretation. The child interviews will be analysed first and separate to that of the adult and professional interview data.

This research will also utilise NVivo in the data analysis, a qualitative software which has been identified as adding validity to qualitative research (Bringer et al., 2004). The data inputted into this software will be the pseudonymised data. Analysis of the data will be conducted on a home-based laptop, that is password protected. Each of the files will be password protected also.

# **PARTICIPANTS**

# **Description of study participants**

# **Child Participants**

Participants of this research will be aged above 16 years old. They will currently be experiencing parental imprisonment.

# **Adult Participants**

This refers to the non-offending parent/career/guardian to the child currently experiencing parental imprisonment.

The participant will above aged 18 years old and the carer/parent/guardian to the child participant.

# **Professional participants**

The professional participant refers to a professional working with the young person or family during parental imprisonment. They will be above 18 years old and currently working with the family during parental imprisonment. This research will aim to recruit a minimum of one child participant and one adult participant.

#### Inclusion criteria

#### **Adult Participant**

- Is the parent/caregiver/guardian to a child (above 16 years old) currently experiencing parental imprisonment
- Participants are based in the UK (England, Wales, Scotland, or Northern Ireland), and have experienced parental imprisonment whilst in the UK.

#### **Child Participant**

- Child participants are above 16 years old at the time of data collection.
- Child participants are currently experiencing parental imprisonment.
- Participants are based in the UK (England, Wales, Scotland, or Northern Ireland), and have experienced
  parental imprisonment whilst in the UK.

#### **Professional Participant**

- Is a professional working with, or previously worked with the family or child impacted by parental imprisonment
- Has worked with the family or child impacted by parental imprisonment for at least one month.
- Participants are based in the UK (England, Wales, Scotland, or Northern Ireland), and have experienced
   parental imprisonment whilst in the UK.

#### **Exclusion criteria**

# **Adult Participant**

- Are the parent of the child participant who was imprisoned.
- Not the current caregiver/guardian/parent to the child participant

# **Child Participant**

- Child participants are the direct victim of their parental offence.
- The child participant is aware of their parent's offence and imprisonment.
- Below 16 years old at the time of data collection.

# **Professional Participant**

• Professional participant is aware that the child's parent is in prison

# Recruitment

Adult and child participants will be recruited through voluntary purposive sampling. The research will be advertised on several social media platforms (including LinkedIn, Twitter, and Reddit), and organisational and charitable websites that work with families of those convicted of offences (including but not limited to Children Heard and Seen, Safer Lives, and Prison Advice Care Trust).

It will be requested that the adult and child participant contacts the lead researcher to volunteer to partake in this research. If the child participant contacts the researcher to participate, it will be requested that they share the research with the adult participant to volunteer to partake. If the adult participant contacts the researcher to participate, it will be requested that they share the research with the child participant to volunteer to partake. It will be requested that both the child and adult participant partake in this research to provide a case study design.

The professional participant will be recruited via opportunity sampling. The non-offending parent/caregiver guardian participant will be encouraged to share the research poster with a professional that works with the family/young person who will then have the option to volunteer to partake in this research.

Verbal and written consent will be collected from all participants researcher via informed consent sheet, and at the interview. After interviews with the participants, all participants will be provided with a debrief and provided with support services to access.

# Screening and eligibility assessment

Participants will be recruited through voluntary purposive sampling. The research will be advertised on several social media platforms (including LinkedIn, Twitter, and Reddit), and organisational and charitable websites that

work with families of those convicted of offences (including Children Heard and Seen, Safer Lives, Prison Advice Care Trust; PACT).

A demographic questionnaire will be administered as a pre-screening assessment at the beginning of the research to ensure that they fit the inclusion and exclusion criteria. If they do not fit the criteria at the time of data collection, they will be directed to exit the research.

Participants will also be provided about information of the research in the preliminary discussions. As part of this, the sensitive nature of this research will be described and explained. If participants feel that they are in a vulnerable place at the time of data collection, and unable to cope with the line of questions in this research, they will be directed to support services and to exit the research.

# Information provided to participants

Participants will be provided with information regarding this research, including the type of questions that will be asked, and aims of the research. First, the research will be advertised using a poster which will outline the aims of the research explicitly, and what type of questions the research might ask.

# **Adult and Child Participant**

Initially, the research will be advertised on online social media platforms and charitable organisations using a poster and a link to express interest in the current research (please see appendices). The poster will include information regarding the title of the research, and it's aims. Participants will be directed to email the researcher, or directed to access a link whereby they will be invited to input their name and email for the researcher to contact them.

Once the participant has contacted the lead researcher, the participant will be provided with an informed consent sheet. Please see appendices. Again, this provides information about the current research. From reading this consent sheet, participants can express interest to participate in the research through contacting the researcher directly via email. Informed consent will be documented by asking for participants to sign the informed consent sheet.

The participant will also have the opportunity to ask any questions they have about the research before deciding to participate within the preliminary discussion, offered to all participants. Within this preliminary discussion the researcher will explain the study, the type of questions and themes which may be asked throughout the interview. A further understanding of the interview and its sensitive nature will be provided.

Participants will further be directed to the researcher's email address if there are any further questions before partaking in the research.

At the start of the scheduled interview, the researcher will read out the informed consent sheet to the participant and ask for the participants understanding of this research. Both written and verbal consent will be sought.

They will also be provided with a debrief of the current research, including their right to withdraw, and information to access support.

#### **Professional participant**

The same information and process as the adult participant will be adhered to with the professional participant. They will also be provided with a debrief of the current research, including their right to withdraw, and information to access support.

#### **Informed Consent**

Informed consent will be obtained on several occasions throughout this research. Informed consent will be sought from all participants prior to, during, and following participating in the current research.

# Participant confidentiality

This research will not store or record any identifiable information.

This study will safeguard the privacy of participants' personal data, and comply with the General Data Protection regulation (GDPR) Data Protection Act 2018, which requires all personal data to be anonymised as soon as it is practical to do so.

Participants are requested to email the research to partake in this research, and thereby the participants name and email address will be known to the researcher. Once the participant has consented to a study, they will be allocated a pseudonym by which they will be referred there forward in documentation. The document of participant information and consent forms will be contained within a password protected file and saved on a password protected home-based computer. Once all participants have been recruited, this file (containing participant information and consent forms) will be removed from the researcher's laptop. For participants that expressed an interest but did not participate (either through choice or being found unsuitable) basic demographic information will be kept in addition for reason for not participating, but all identifiable information (such as name and contact details) will be deleted.

The interviews will be conducted via Microsoft Teams and will be audio recorded using this function on Teams. The interviews will also be transcribed live using the online transcribing feature of Teams. This will be on a password protected laptop. The audio file will be password protected and saved as the pseudonym which was allocated to them following consent. Once the interview has been completed, the researcher will go through the recording and transcription to ensure that they are congruent. The transcription document will be password protected saved also, and stored securely on password protected device. During transcription, any identifiable information will be pseudonymised whereby they will be changed to their assigned pseudonym. Pseudonyms will be used in replacement of any identifiable information.

This research will also utilise NVivo in the data analysis, a qualitative software which has been identified as adding validity to qualitative research (bringer et al., 2004). The data inputted into this software will be the pseudonymised formatted transcribed data.

This research cannot be completely anonymous as in the dissemination of findings, direct quotes may be taken from the pseudonymised interviews. However, any information included will not be identifiable to an individual (including

their name, geographical place etc). Furthermore, any direct quotes used will focus on their experiences rather than the individual themselves, and this will be referred to using a generated pseudonymised name.

It is also worth noting that what is discussed in each individual interview, will not be shared with any other participants that partake in this research. At the beginning of interviews with participants, it will be explained that any information that is disclosed during the interview that would suggest a risk of harm to themselves, or another person will need to be disclosed to the appropriate persons (e.g. Police, Local Safeguarding Teams, 111, or the parent if disclosed by the child).

#### Incentive

At the end of completing the qualitative and quantitative data, participants will be invited to voluntarily provide their email address to enter a raffle to win a voucher of £15 (one of four vouchers) for their participation. Participants' email addresses will be stored in a file stored separately to data collected for this research. This file will be password protected. Following data collection, the raffle will be run and the winning participants will be contacted via email to provide the gift card. All emails will then be deleted and destroyed from the computer systems.

# Discontinuation/ withdrawal of participants from study

Participants will be able to withdraw from the study at any point prior to attending interview with the lead researcher. Their right to withdraw from the study will be and/or can be without reason. Participants will be informed of their right to withdraw in the informed consent sheet, during preliminary discussion, and during the interview.

Following the interview, participants will be provided with a debrief. It will be outlined that participants can withdraw from their involvement in the current study up to two weeks after partaking in this research without needing a reason. Once two weeks (14 days) from the day of interview have passed, participants will be unable to withdraw from this study. Participants will be informed of this.

# Definition of end of study

#### Adult participant

The end of participant involvement will be after the adult and child interview with the lead researcher has finished.

# **Child participant**

The end of participant involvement will be after the interview with the lead researcher has finished.

# **Professional participant**

The end of participant involvement will be after the interview with the lead researcher has finished.

**Expenses and benefits** 

Not applicable.

# ETHICAL CONSIDERATIONS AND PARTICIPANT AND RESEARCHER SAFETY

Most research carries the risk of some ethical challenge. If this is the case, you need to demonstrate your awareness of the problem and your response to mitigate ethical objections. There is a free text box below to detail any study specific ethical issues, however the following areas are often a cause for concern:

| Please indicate which of the below criteria apply to your project. | | |
|---|---|---|
| | Yes | No |
| Research projects that give rise to evident and significant risk of reputational damage to, or legal liability | | Х |
| on the part of, the Researcher or the University of Nottingham. | | ^ |
| | | I |
| Procedures where the probability and magnitude of harm or discomfort anticipated in the research | | |
| project are greater in and beyond those ordinarily encountered in daily life or during the performance | | Х |
| of routine physical or psychological examinations or tests. | | |
| Procedures the nature of which might be offensive, distressing or deeply personal for the target group. | Х | |
| This may include surveys and questionnaire-only research designs. | | |
| The research may be personal for participants as it asks participants to share their experiences of paren | ntal | |
| imprisonment. The research has aimed to reduced the anticipated distress experienced by the participa | ant by | |
| providing information about the true aims and content of the research. | | |
| Research projects that involve children under the age of 16 or other vulnerable groups. | Х | |
| This research aims to recruit child aged 16 years or above who currently have a parent in prison. It will also aim to | | m to |
| recruit the non-offending parent, caregiver, or guardian to the child, and a professional working with the family or | | |
| child participant. The available evidence base suggests that the experience of parental imprisonment may expose | | |
| an individual to adverse experiences and several collateral consequences, thereby making this a vulnerable | | |
| population. | | |
| The child participant will be offered to complete the interview in the presence of the adult participant. | | |
| Research projects involving prisoners or young offenders. | | Х |
| Research projects involving police, probation services, or those involved in the criminal justice system. | | Х |

| Research projects that involve those who may feel under pressure to take part due to their connection | | |
|---|---|---|
| with the researcher (e.g. PI asking their students to participate in their research project or a researcher | | Х |
| asking the people they manage to take part in their research). | | |
| Research designs requiring participants to take part in the research project without their knowledge | | |
| and/or consent at the time and research projects that involve deception or withholding information from | | Х |
| research participants even if the research participants are briefed afterwards. | | |
| Research projects accessing records and/or the collection of personal data, concerning identifiable | | Х |
| individuals as defined by data protection legislation. | | |
| Research projects involving the linking or sharing of personal data, special category data (Sensitive | | Х |
| data) or confidential information beyond the initial consent given. | | |
| Research projects involving the collection or access of audio, video recordings, photographs or | | |
| quotations where individuals may be identified (beyond images that are in the public domain and are | X | |
| being used in their intended context e.g. photographs of politicians). | | |
| It is important to note that the dissemination of findings is expected to include quotations from the qualitative story | | |
| stem data. However, this will be in pseudonymised format (any information included will not be identifiable to the | | |
| individual including their name, geographical place etc) and will only focus on their narratives and experiences. | | |
| Research projects offering incentives which may unduly influence participants' decision to participate. | Χ | |
| Participation in this research study will be incentivised with the chance to win one of four £15 Love2Shop | | |
| vouchers. This will be advertised to participants on the posters and leaflets created. At the end of completing the | | the |
| qualitative and quantitative data, participants will be invited to voluntarily provide their email address to | qualitative and quantitative data, participants will be invited to voluntarily provide their email address to enter a | |
| raffle to win a voucher for their participation. This incentive may influence a participants' decision to participate in | | te in |
| the current study, however, it is optional to enter the raffle. Participants will also be asked to provide their email | | ail |
| address at the end of research completion to reduce any potential undue influence. | | |
| Research projects that are likely to lead to incidental findings or disclosures. | | Х |
| Research projects carried out by third parties wishing to recruit University of Nottingham's staff and/or | | Х |
| students as participants | | |
| Research projects involving the new collection or donation of human tissue from a living person or the | | Х |
| recently deceased as defined by the Human Tissue Authority (HTA). | | |

| Research projects which had previously received a favourable ethical opinion (FEO) but had not | Х |
|---|---|
| started within a year of the FEO. | |
| Research projects which had previously received an FEO but have not been completed within five | X |
| years of the FEO date. | |
| Research projects involving <b>travelling</b> to countries/regions <b>against</b> the advice of the British Foreign | Х |
| Commonwealth Office. | |
| Research Projects involving data collection outside the UK (except at UoN international campuses). | X |
| Research projects involving activities or the outcome of which may pose a security risk or may be perceived to pose a security risk. i.e. Counter-Terrorism and Security Act (Prevent Duty guidance), | X |
| which seeks to prevent people from being drawn into terrorism? | |
| The state of the s | |
| Decouple projects in relating activities that acrid natarities, appropriate the activities of the | |
| Research projects involving activities that could potentially compromise the safety/wellbeing of the researcher. | X |
| Please give details of any other study-specific ethical and/or safety considerations | |
| Additional Checks: | |
| Additional Offices. | |
| Does the research involve fieldwork or data collection off campus? | |
| □ Yes ⊠ No | |
| If we where confirm that a Diela Accomment has been completed and signed off by the annuari | oto Cofoty |
| If yes, please confirm that a Risk Assessment has been completed and signed off by the appropria Officer/Supervisor. | ile Salety |
| Is the research project going to be conducted outside the UK or involves international partners? | |
| □ Voo □ № No | |
| ☐ Yes ☐ No | |

| Please confirm all relevant permissions (including where applicable Non-UK REC approval/Favourable |
|---|
| Ethical Opinion) have been or will be in place before the relevant research activities commence. |
| □ I confirm |

# **DATA MANAGEMENT SUMMARY**

| William III have a second of the second of t | |
|---|---|
| Who will have access to the <u>research</u> data? | The primary researcher (Kyra Wardle, DForenPsy Student) |
| | and supervising researcher (Dr Elizabeth Paddock) will have |
| | access to the data. The research supervisor will have access to |
| | the data over the University of Nottingham secure server. |
| | Direct access will be granted to authorised representatives |
| | from the University of Nottingham and any host institution for |
| | monitoring and/or audit of the study to ensure compliance |
| | with regulations. |
| How will <u>research</u> data be stored? | The research will be stored on a password protected home- |
| | based laptop, and also be password protected. |
| | The data collected from participants will be stored securely on |
| | a home-based password protected laptop. These file names |
| | will be saved as the participant number provided to each |
| | participant so that this is not identifiable, and will also be |
| | password protected. |
| | As this research utilises semi-structured interviews, it is |
| | possible that the participant will share identifiable personal |
| | information during the interview. If the qualitative data |
| | includes any identifiable or personal information, this will be |
| | pseudonymised immediately following the interview. The |
| | pseudonymised data will be stored securely on a password |
| | protected device, and the document itself will be password |
| | protected and saved as the participant's number. The |
| | identifiable qualitative information will be destroyed as soon |
| | as this is pseudonymised. |
| | as this is pseudonymised. |

| | At the end of completing the qualitative and quantitative |
|---|---|
| | data, participants will be invited to voluntarily provide their |
| | email address to enter a raffle to win a voucher for their |
| | participation. Participants' email addresses will be stored in a |
| | file stored separately to data collected for this research. Their |
| | email address will be stored separately to their unique |
| | identification number and data collected as part of this |
| | research. This file will also be password protected. Following |
| | data collection, the raffle will be ran and the winning |
| | participants will be contacted via email to provide the gift |
| | card. All emails will then be deleted and destroyed from the |
| | computer. |
| How long will <u>research</u> data be stored for? | The data will be stored for the minimum retention period of 7 |
| | years following the end of the study, in line with the University |
| | of Nottingham's retention period requirements. |
| What will be done with the <u>research</u> data at the | At the end of the storage period, the research data will be |
| end of the storage period? | destroyed and deleted. |
| Who will have access to the participants' | The primary researcher (Kyra Wardle, DForenPsy Student) |
| personal data? | |
| How will <u>personal</u> data be stored? | The data collected from participants will be stored securely on |
| | a home-based password protected laptop. These file names |
| | will be saved as the participant number provided to each |
| | participant so that this is not identifiable. These files will also |
| | be password protected. |
| | As this research utilises online survey methods, no identifiable |
| | information will be stored. Participants' demographic |
| | information and qualitative data will be saved as their |
| | participant number. |
| How long will <i>personal</i> data be stored for? | To comply with the Data Protection Act, personal data will be |
| | deleted as soon as possible after it is no longer needed for the |
| | study. |
| Describe method(s) of research data | All demographic data will be entered on an Excel spreadsheet. |
| entry/management | The participants will be identified by a unique study specific |
| | number and/or code in any database. Their name or any |

other identifying detail will NOT be included in any study data electronic file.

Qualitative data will be stored on NVivo for analysis. Only the pseudonymised transcripts will be uploaded to NVivo for analysis. The participants will be identified by a unique study specific number and/or code in any database. Their name or any other identifying detail will NOT be included in any study data electronic file.

# STUDY MONITORING AND OVERSIGHT

# Who will be responsible for day-to-day supervision of the study?

Primary Researcher (Kyra Wardle, DForenPsy Student)

Give information about frequency of meetings that will be held to discuss progress/problems. Who will be present at the meetings?

The primary researcher (Kyra Wardle, DForenPsy Student) and research supervisor (Dr Elizabeth Paddock) will meet on a monthly basis to discuss progress and any problems with the current research project.

#### ETHICAL AND REGULATORY CONSIDERATIONS

# **Declaration of Helsinki**

The PI will ensure that this study is conducted in accordance with the principles of the Declaration of Helsinki.

# Research Ethics review and favourable opinion

This form, an informed consent form, a participant information sheet(s) and any proposed advertising material will be submitted to the UoN FMHS REC for written Favourable ethics Opinion (FEO). The research team will submit and, where necessary, obtain approval from the UoN FMHS REC and any other above-mentioned parties for all amendments to the original documents given an FEO.

# **End-of-Study Report**

The PI shall request, complete and submit an end-of-study report to the UoN FMHS REC within 6 months of the study end (participant involvement).

# **INSURANCE AND INDEMNITY**

Insurance and indemnity for University employees, its agents and students conducting University business is provided through several policies and will respond in the event of a successful litigious claim for proven negligent harm.

#### **DISSEMINATION AND FEEDBACK OF STUDY OUTCOMES**

The results of this research will be disseminated as a DForenPsy Research Thesis and be considered for publication. The results of this research will also be shared with a Viva panel board, as part of the requirements of this course.

As this research will utilise the support of Charitable Organisations for the recruitment of participants, if requested, the final research thesis will be shared with them.

# **REFERENCES**

- Aebi, M., & Cocco, E. (2023). Map 1. Prison population rates (number of inmates per 100,000 inhabitants) on. 31
- Barnardo's (2016) Children of prisoners. A guide for community health professionals [online]. Essex: Barnardo's.

  Available from: https://www.nicco.org.uk/userfiles/downloads/5ae18e3dd0bb4-767-i-hophealth-guide.pdf
- Beresford, S., Loucks, N., & Raikes, B. (2020). The health impact on children affected by parental imprisonment. *BMJ paediatrics open*, *4*(1), e000275.
- Bowlby, J. (1973). Attachment and Loss
- Braun, V., & Clarke, V. (2006, January). *Using thematic analysis in psychology*. Qualitative Research in Psychology.
- Braun, V., Clarke, V., Hayfield, N., Frith, H., Malson, H., Moller, N., & Shah-Beckley, I. (2019). Qualitative story completion: Possibilities and potential pitfalls. *Qualitative Research in Psychology, 16*(1), 136–155.
- Bringer, J. D., Johnston, L. H., & Brackenridge, C. H. (2004). Maximizing Transparency in a Doctoral Thesis1: The Complexities of Writing About the Use of QSR\*NVIVO Within a Grounded Theory Study. *Qualitative Research*, 4(2), 247–265. https://doi.org/10.1177/1468794104044434
- Bülow, W. 2014. "The Harms beyond Imprisonment: Do We Have Special Moral Obligations towards the Families and Children of Prisoners?." Ethical Theory and Moral Practice 17 (4): 775–89.
- Clarke, V., & Braun, V. (2013, March). Successful qualitative research: A practical guide for beginners.

  ResearchGate: Sage.
- Clarke, V., Hayfield, N., Moller, N., Tischner, I., & undefined, undefined. (2017). *Once Upon a Time ...: Qualitative Story Completion Methods* (D. Gray, V. Clarke, & V. Braun, Eds.). Cambridge University Press; Cambridge University Press.
- Dobbie, W., H. Grönqvist, S. Niknami, M. Palme, and M. Priks. 2019. The Intergenerational Effects of Parental Incarceration. Institute for Evaluation of Labour Market and Education Policy. Working Paper 2019: 24.
- Felitti, V. J., Anda, R. F., Nordenberg, D., Williamson, D. F., Spitz, A. M., Edwards, V., Koss, M. P., & Marks, J. S. (1998). Relationship of Childhood Abuse and Household Dysfunction to Many of the Leading Causes of Death in Adults. *American Journal of Preventive Medicine*, 14(4), 245–258.

- Gavin, H. (2005). *The Social Construction of the Child Sex Offender Explored by Narrative*. <a href="https://eprints.hud.ac.uk/id/eprint/9504/1/gavin.pdf">https://eprints.hud.ac.uk/id/eprint/9504/1/gavin.pdf</a>
- Jaffee S, Moffitt T, Caspi A, Taylor A. "Life With (or Without) Father: The Benefits of Living With Two Biological Parents Dependent on the Father's Antisocial Behavior" *Child Development*. 2003;74:109–26
- Lam, L., & Comay, J. (2020). Using a Story Completion Task to Elicit Young children's Subjective Well-Being at School. *Child Indicators Research*.
- Lotto, L. S., Miles, M. B., & Huberman, A. M. (1986). Qualitative Data Analysis: A Sourcebook of New Methods. *Educational Evaluation and Policy Analysis*, 8(3), 329.
- Lowenstein, Ariela. (1986). Temporary Single Parenthood--The Case of Prisoners' Families. Family Relations. 35. 10.2307/584286.
- Manby, M., Jones, A. D., Foca, L., Bieganski, J., & Starke, S. (2014). Children of prisoners: exploring the impact of families' reappraisal of the role and status of the imprisoned parent on children's coping strategies. *European Journal of Social Work*, 18(2), 228–245.
- McGinley, M. and Jones, C. (2018) Growing Up with Parental Imprisonment: Children's Experiences of Managing Stigma, Secrecy and Shame. Practice [online]. 30 (5), pp. 341-357
- Moller, Naomi & Clarke, Victoria & Braun, Virginia & Tischner, Irmgard & Vossler, Andreas. (2021). Qualitative Story Completion for Counseling Psychology Research: A Creative Method to Interrogate Dominant Discourses. Journal of Counseling Psychology.
- Moore, S. M., Gullone, E., & Kostanski, M. (1997). An examination of adolescent risk-taking using a story completion task. *Journal of Adolescence*, *20*(4), 369–379.
- Murray, J., & Farrington, D. (2008a). The Effects of Parental Imprisonment on Children.
- Murray, J., & Farrington, D. P. (2008b). PROTOCOL: Parental Imprisonment: A systematic review of its effects on child antisocial behavior, crime and mental health. *Campbell Systematic Reviews*, 4(1), 1–44.
- Oppenheim, D., Emde, R. N., Hasson, M., & Warren, S. (1997). Preschoolers face moral dilemmas: A longitudinal study of ackowledging and resolving internal conflict. *International Journal of Psycho-Analysis*, 9(1), 1–9.
- Reeves, C. (2016) Experiencing imprisonment: research on the experience of living and working in carceral institutions [online]. London: Routledge.
- World Health Organization. (2020, January 28). Adverse Childhood Experiences International Questionnaire (ACE-IQ).

#### **DECLARATIONS AND SIGNATURES**

# I/We, the researcher(s):

- Understand our responsibilities in line the University of Nottingham Code of Research Conduct and Research Ethics and UoN Policies and Guidance
- Understand that, for studies conducted outside the UK, it is my/our responsibility to understand and adhere to all local regulations and guidelines and will ensure all required permissions are in place before any relevant Research activities commence
- The research project activities will not commence before obtaining favourable ethical opinion from FMHS REC and any other relevant permissions
- Understand the Principal Investigator must ensure all researchers are suitably qualified and trained to conduct the research described, or are appropriately supervised until deemed qualified/trained
- Agree to maintain the confidentiality of the research participants and will grant access to data only to authorised persons.
- Agree to immediately notify the REC in writing of any proposed change to the research as outlined in this application and await approval before proceeding with the proposed change

- Make arrangement to stop the research project if the Principal Investigator changes and notify the REC of the successor
- · Will use the data collected only for the purposes outlined in this application and participants have consented to
- Have made arrangements to ensure that <u>personal data</u> collected from participants will be held in compliance with the requirements of the GDPR and the Data Protection Act 2018.

#### **Useful links:**

- 1. Code of Research Conduct and Research Ethics
- Reading the following Code of Practice for Research Ethics Committees should give you a clear understanding of the review criteria used to assess research projects and help you plan your study. <u>Code</u> of Practice for Research Ethics Committees
- 3. UKRIO Recommended Checklist for Researchers
- 4. Access and Benefits Sharing and Nagoya Protocol
- 5. UoN Information Security and Compliance Team for advice on using personal data and GDPR <a href="https://uniofnottm.sharepoint.com/sites/InformationSecurityandCompliance/">https://uniofnottm.sharepoint.com/sites/InformationSecurityandCompliance/</a>
- 6. Research Misconduct
- 7. International Research and Research Ethics Research Conduct in an International context
- 8. Research Integrity Bytes: one pagers addressing common issues and questions raised by researchers in all fields. The bytes are written to give researchers a starting point when considering issues that may impact the integrity of their research.
- Research projects involving NHS patients and/or staff and/or their data: see the <u>Research Governance</u> workspace pages
- 10. <u>UoN Safeguarding Resources</u> a plan needs to be in place if something of concern is likely to be raised
- 11. Create a secure online survey
  <a href="https://uniofnottm.sharepoint.com/sites/DigitalResearch/SitePages/Surveys.aspx">https://uniofnottm.sharepoint.com/sites/DigitalResearch/SitePages/Surveys.aspx</a>
- 12. Automated Transcription Service https://uniofnottm.sharepoint.com/sites/DigitalResearch/SitePages/Automated-Transcription.aspx
- Cyber Essentials Secure SharePoint
   https://uniofnottm.sharepoint.com/sites/DigitalResearch/SitePages/Secure-SharePoint--Cyber-Essentials.aspx
- 14. Digital Research Planning, Data storage, Process & analyse, Promote & archive.
- 15. Insurance Team: https://uniofnottm.sharepoint.com/sites/Insurance2

# **Check List**

- Data management Plan (your application cannot be reviewed without one)
- Participant Information Sheet
- Consent Form
- Poster, invite e-mails, draft of text to be used in social media- note: monetary amounts should not be stated
- Letters of permission from gatekeepers, outside institutions, where applicable
- Copy of proposed questionnaire and web link if online where applicable
- Outline of interviews or focus group discussions including online material instructions where applicable
- Plan of action in case there is a problem or something of concern is raised.
- Demographic questionnaires or other relevant additional materials where applicable
- For Research being conducted overseas: an outline of the research ethics regulations, local laws and permissions required. Cultural setting and context should be included in the section of the form
- Any additional relevant information i.e., translations into other languages, large print for visually impaired

Please submit form and supporting documents by e-mail as attachments to:

FMHS-ResearchEthics@nottingham.ac.uk